CLINICAL TRIAL: NCT04963998
Title: Safety and Efficacy Study of MedCu Wound Dressings With Copper Oxide
Brief Title: Safety and Efficacy Study of MedCu Wound Dressings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MedCu Technologies Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WD-2C-1010-01-IL
Record Dates: First submitted 2021-06-28; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Wounds and Injuries; Diabetes Complications
Keywords: wound dressings; copper oxide; diabetic ulcers
MeSH Terms: conditions — Wounds and Injuries; Diabetes Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Copper oxide dressings (Experimental): Treatment of diabetic ulcers that were in a stagnated stage with copper oxide containing wound dressings
  Interventions: Device: Application of Wound Dressings with Copper Oxide

INTERVENTIONS:
Device: Application of Wound Dressings with Copper Oxide — Application of Wound Dressings with Copper Oxide on chronic foot wounds in diabetic patients

SUMMARY:
The Study was divided into three Phases: Screening Phase (1-2 weeks); Treatment Phase (~ 1 month); and Follow-up Phase (two weeks). During the Screening Phase, blood samples were taken for analysis of blood count, liver and kidney functions from potential appropriate diabetic patients with chronic wounds in their foot. Stable chronic diabetic patients, whose wounds were not infected and the wound size increased or did not decreased by more than 25% per week or 35% by SOC treatment during the Screening Phase, and who will meet all other study inclusion criteria, were enrolled and start the 4 weeks Treatment Phase. The wounds were then treated by applying the Copper Oxide containing Dressings (COD) that were changed twice a week. In the two weeks post-treatment period, the patient received standard of care (SOC) dressing. In that time period, the patient were seen once after two weeks. The Primary outcome was the evaluation of the safety of the COD and the secondary outcomes were the evaluation of the wound size change of the foot wounds when using COD. Measures that were assessed included

1. Percent change in wound size during the Treatment Phase,
2. Rate of increase in extent and quality (color) of granulation tissue,
3. Infectious episodes during the Treatment Phase.

DETAILED DESCRIPTION:
The Study was divided into three Phases: Screening Phase (1-2 weeks); Treatment Phase (~ 1 month); and Follow-up Phase (two weeks). During the Screening Phase, blood samples were taken for analysis of blood count, liver and kidney functions from potential appropriate diabetic patients with chronic wounds in their foot. Stable chronic diabetic patients, whose wounds were not infected and the wound size increased or did not decreased by more than 25% per week or 35% by SOC treatment during the Screening Phase, and who will meet all other study inclusion criteria, were enrolled and start the 4 weeks Treatment Phase.

During the Treatment Phase, the index wounds were evaluated, undergone bed side debridement if necessary, and photographed. Tissue Analytics software was used to assess wound size and volume. The wounds were washed by normal saline or a previously used solution (but no new disinfectant or any antibacterial preparation), and then the COD was applied on the wound. The COD was applied on the wounds for the duration of the Treatment Phase and changed twice a week, once in the clinic and once at home. At every clinic visit the following assessments were performed: wound assessment, including size determination, depth, clinical impression of infection (swelling, erythema, discharge quantity and quality, granulation, fibrin and necrotic tissue, odor, pain, and tenderness); antibiotics and vital signs as necessary. After ~ 1 month of test wound dressings use, a blood sample was taken for blood count, liver and kidney functions. If needed, the patients' wounds were treated using the hospital SOC in the follow up period. The Primary outcome was the evaluation of the safety of the COD and the secondary outcomes were the evaluation of the wound size change of the foot wounds when using COD. Measures that were assessed included

1. Percent change in wound size during the Treatment Phase,
2. Rate of increase in extent and quality (color) of granulation tissue,
3. Infectious episodes during the Treatment Phase.

ELIGIBILITY:
Inclusion Criteria:

Patients must satisfy all of the following inclusion criteria to be included in the study:

1. Male or female subjects, 18 to 80 years of age at the time of enrollment.
2. Subject has Diabetes Mellitus (type 1 or type 2) by WHO criteria.
3. Wound exists for at least 4 weeks including 4 weeks from last surgical debridement in operating room (OR) or minor foot amputation.
4. The foot wound size has not decreased by more than 25% per week or 35% in two weeks by SOC during the screening period.
5. Wound size 2-30 cm2.
6. The wound does not have signs of infection as defined by Dumville et al., Topical antimicrobial agents for treating foot wounds in people with diabetes. Cochrane Database of Systematic Reviews 2017, Issue 6. Art. No.: CD011038, Table 1. For clarity, the following signs are allowed:

   1. If erythema is present at wound it should be up to 2 cm from the wound edges.
   2. If exudate is present it should be either serous or thick but not thick-purulent nor purulent
   3. Green or black necrotic tissue constitute up to 20% of the wound size.
7. The wound should not have cavities or deep sinuses. However, cover by free skin or soft tissue wall is allowed for up to 5 mm.
8. Having at least moderate blood perfusion into the affected limb as defined by palpable pulses (Dorsalis Pedis and/or Tibialis Posterior, unequivocally palpable). If no pulse is clearly present in vascular lab tests Ankle Brachial Index (ABI) should be 0.6< or if ABI > 1.3, then toe pressure of > 50 mmHg.
9. Having a body mass index (BMI) <40 Kg/m2.
10. Recent glycosylated haemoglobin (HbA1c) <12.0%.
11. Not undergoing any systemic or topical antibiotic treatment for the wound for a week before enrollment in the study.
12. No foot deformity or bony projection that is severe enough to jeopardize wound healing as deemed to the treating physician.
13. The patient is able and eligible to sign written informed consent and participate in the study.
14. Be available for the entire study period, and ability and willingness to adhere to the requirements of the study.

Exclusion Criteria:

Patients will be excluded from the study if they meet any of the following exclusion criteria:

1. General conditions:

   * A clinically significant active or unstable cardiac, gastrointestinal, endocrine, neurological, liver, or kidney disease.
   * Psychiatric condition.
   * Active participation in an investigational trial within 30 days of the screening visit.
   * History of allergic reactions attributed to copper.
   * Subjects with Active Charcot neuro-arthropathy.
   * Any chronic or acute condition susceptible of interfering with the evaluation of the wound dressing effect.
   * Individuals using and need to continue use any type of topical agents in or on the wound.
   * Any form of substance abuse (including drug or alcohol abuse, excluding cannabis), psychiatric disorder or any chronic condition susceptible, in the opinion of the investigator, of interfering with the conduct of the study.
   * Females who are pregnant, lactating, of child-bearing potential.
   * Fertile female subjects who are not willing to use an acceptable method of contraception during the treatment period and for 14 days following completion of treatment.
   * Subjects who are likely to be non-compliant or uncooperative during the study.
2. Laboratory tests:

   * Anemia (Hemoglobin < 8.0 g/dL).
   * White Blood Cells count > 11,000/μL.
   * Platelets count < 100,000/μL.
   * Liver function tests > 3 times upper normal lab values.
   * Creatinine > 3.5 mg/dL.
   * Albumin < 2.2g/dL.
   * Any other clinically significant blood and urinalysis tests abnormalities that can jeopardize study results as evaluated by the investigator.
3. Wound condition:

   * The wound size area has decreased by more than 25% per week or 35% in two weeks by SOC treatment during the screening phase prior to the commencement of the study.
   * Have visible bone exposed at wound site.
   * Any signs of infection in the wound (which could be linked to raised body temperature), abscess, cellulitis, necrosis, drainage or known osteomyelitis or erythema around the wound of more than 2 cm.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2020-10-21 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 4 weeks
  Incidence of Treatment-Emergent Adverse Events as assessed by determination
  * Vital signs
  * Physical Examination of the treated wound
  * Sensitivity to the wound dressing
  * Complete Blood Tests, which include complete blood counts (CBC), Liver and Kidney Function tests, and C-reactive protein (CRP)
  * Concomitant medication use.

SECONDARY OUTCOMES:
Percent change in wound size | 4 weeks
  The percent of wound size of the foot wounds when using Wound Dressings with Copper Oxide (COD) was determined by using Tissue Analytics 3D Wound Imaging System. At each time point the size of the wound was compared to the initial size of the wound when starting using the COD.
Rate of change in extent and quality (color) of granulation tissue | 4 weeks
  The extent and quality of the color of the wound tissue was assessed by using both the Tissue Analytics 3D Wound Imaging System and physicians clinical evaluation. The percent of the granulation tissue at each time point was compared to the initial quality of the granulation tissue at the beginning of the treatment with the COD.
Rate of change in percent of fibrin tissue | 4 weeks
  The percent of change in the percent of fibrin tissue was analyzed the Tissue Analytics 3D Wound Imaging System and by the physicians clinical evaluation. The percent of the fibrin tissue at each time point was compared to the initial percent of the fibrin tissue at the beginning of the treatment with the COD.

CONTACTS AND LOCATIONS:
Overall Officials: Alexei Rovitsky, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No